CLINICAL TRIAL: NCT02934607
Title: A Randomised, Open-Label, Single-Dose, Single-Centre, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of Symbicort pMDI 160/4.5µg Administered With a Spacer (With and Without Charcoal) and Symbicort pMDI 160/4.5µg Administered Without a Spacer (With and Without Charcoal)
Brief Title: A Study to Assess How Much Drug Reaches the Blood When Given From Symbicort pMDI With Spacer Compared to That of Symbicort pMDI Without Spacer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D589WC00001; 2016-001866-27 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-10-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Study is Being Conducted in Healthy Volunteers
Keywords: Asthma; Chronic obstructive pulmonary disease; Spacer device; Symbicort; Pressurized metered-dose inhaler; Relative bioavailability; Crossover; AstraZeneca; Safety; Activated charcoal; AeroChamber Plus Flow-Vu spacer device
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Anthrax | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): 2 x 160/4.5 µg Symbicort pMDI administered with no spacer device; no activated charcoal (systemic exposure).
  Interventions: Drug: Symbicort pMDI without spacer device
- Treatment B (Experimental): 2 x 160/4.5 µg Symbicort pMDI administered through AeroChamber Plus Flow-Vu spacer device; no activated charcoal (systemic exposure).
  Interventions: Drug: Symbicort pMDI with spacer device
- Treatment C (Active Comparator): 160/4.5 µg Symbicort pMDI administered with no spacer device; with activated charcoal (lung exposure).
  Interventions: Drug: Symbicort pMDI without spacer device
- Treatment D (Experimental): 160/4.5 µg Symbicort pMDI administered through AeroChamber Plus Flow-Vu spacer device; with activated charcoal (lung exposure).
  Interventions: Drug: Symbicort pMDI with spacer device

INTERVENTIONS:
Drug: Symbicort pMDI with spacer device — Relative bioavailability of budesonide and formoterol delivered via Symbicort pressurized metered-dose inhaler (pMDI) with a spacer device (test)
  Arms: Treatment B; Treatment D
Drug: Symbicort pMDI without spacer device — Relative bioavailability of budesonide and formoterol delivered via Symbicort pMDI without a spacer device (reference)
  Arms: Treatment A; Treatment C

SUMMARY:
This study will be conducted to establish the relative bioavailability of budesonide and formoterol delivered via Symbicort pressurized metered-dose inhaler (pMDI) with and without a spacer device.

Administration under each condition will occur with the concomitant administration of activated charcoal to estimate exposure through the lung and without activated charcoal to estimate total systemic exposure.

DETAILED DESCRIPTION:
Study Design:

This study will be a randomised, open-label, single-dose, crossover study in healthy subjects (males and females), performed at a single study centre.

The study will comprise:

* A screening period of maximum 28 days;
* Four treatment periods during which subjects will be resident from the afternoon before dosing with Symbicort until at least 24 hours after dosing; discharged on the morning of Day 2; and
* A final visit within 5 to 7 days after the last administration of Symbicort. There will be a minimum washout period of 3 days between each dose administration of Symbicort. Subjects will receive single doses of Symbicort on 4 occasions under fasted conditions. During screening, spirometry testing will be performed by a technologist or a qualified designee to ensure subjects perform adequate manoeuvres to achieve optimal lung function. Device and inhalation training will be conducted on admission to each treatment period, and prior to dosing on Day 1 of each treatment period.

Duration:

Approximately 7 weeks

Statistical Analysis:

* For total systemic exposure: Treatment B versus Treatment A
* For lung exposure: Treatment D versus Treatment C Treatment ratio will be assessed on the ratio of log-transformed Cmax, AUC0-t and AUC of budesonide and formoterol using a 2-sided 90% confidence interval (CI) approach based on a repeated measures analysis of variance (ANOVA) model including period and treatment as fixed effects, and subject as a random effect. The estimated treatment differences and the 90% CIs on the log scale will be back-transformed to obtain the Gmean ratios for each pair of treatments. The least squares means (and 95% CIs), Gmean ratios and 90% CIs will be tabulated for each comparison and analyte (budesonide and formoterol).

Sample Size:

The sample size is 56 to ensure adequate number of subjects are randomised and at least 44 evaluable subjects complete the study.

Assuming an intra-subject coefficient of variation (CV) of 33% (based on the variability of AUC0-12 for budesonide and AUC0-12 and Cmax for formoterol observed in a similarly designed crossover study in healthy adults), 44 evaluable subjects will give at least 80% power to show that the 90% CI for the treatment effects lies entirely within the range 0.8 to 1.25, i.e., would rule out a 20% change (on a log scale) in exposure to budesonide and formoterol.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 years (inclusive) and older, with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on first admission to the unit, must not be lactating.
4. Body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted value and FEV1/Forced vital capacity (FVC) ratio ≥ 70%.
6. Non-smokers.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History of diagnosed COPD or asthma. (Note: Subjects with a history of childhood asthma only will not be excluded from the study).
3. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
5. Any clinically significant abnormalities in clinical chemistry, 12-lead electrocardiogram (ECG) at screening, haematology, or urinalysis results at screening or vital signs at screening and first admission to the study unit.
6. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody.
7. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
8. Participation in another clinical study with a non-biologic investigational product or new formulation of a marketed non-biologic drug within 3 months prior to the screening visit.
9. Participation in another clinical trial with any marketed or investigational biologic within 4 months or 5 half-lives whichever is longer, prior to the screening visit.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
11. History of severe or ongoing allergy/hypersensitivity (e.g., food allergy) or history of hypersensitivity to drugs with a similar chemical structure or class to Symbicort.
12. Positive screen for drugs of abuse, alcohol or cotinine at screening and on first admission to the study unit.
13. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
14. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. (Note: Hormonal contraception and hormonal replacement therapy are allowed for females, as applicable).
15. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
16. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
17. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Symbicort pMDI administered with spacer device without charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess Cmax of Symbicort pMDI administered through a spacer device without charcoal under fasted condition (total systemic exposure).
  The analysis was done on pharmacokinetic analysis set.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) of Symbicort pMDI administered with spacer device without charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess AUC0-t of Symbicort pMDI administered through a spacer device without charcoal under fasted condition (total systemic exposure).
  The analysis was done on pharmacokinetic analysis set.
Cmax of Symbicort pMDI administered with spacer device with charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess Cmax of Symbicort pMDI administered through a spacer device with charcoal under fasted condition (lung exposure).
  The analysis was done on pharmacokinetic analysis set.
AUC0-t of Symbicort pMDI administered with spacer device with charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess AUC0-t of Symbicort pMDI administered through a spacer device with charcoal under fasted condition (lung exposure).
  The analysis was done on pharmacokinetic analysis set.
Cmax of Symbicort pMDI administered without spacer device without charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess Cmax of Symbicort pMDI administered without a spacer device without charcoal under fasted condition (total systemic exposure).
  The analysis was done on pharmacokinetic analysis set.
AUC0-t of Symbicort pMDI administered without spacer device without charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess AUC0-t of Symbicort pMDI administered without a spacer device without charcoal under fasted condition (total systemic exposure).
  The analysis was done on pharmacokinetic analysis set.
Cmax of Symbicort pMDI administered without spacer device with charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess Cmax of Symbicort pMDI administered without a spacer device with charcoal under fasted condition (lung exposure).
  The analysis was done on pharmacokinetic analysis set.
AUC0-t of Symbicort pMDI administered without spacer device with charcoal | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To assess AUC0-t of Symbicort pMDI administered without a spacer device with charcoal under fasted condition (lung exposure).
  The analysis was done on pharmacokinetic analysis set.

SECONDARY OUTCOMES:
AUC after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the AUC after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Tmax after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the tmax after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½,λz) after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the t½,λz after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Apparent volume of distribution during the terminal phase (extravascular administration) (Vz/F) after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the Vz/F after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the CL/F after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Time of last quantifiable plasma concentration (tlast) after single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the tlast after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Terminal elimination rate constant (λz) after single doses of budesonide and formoterol delivered via Symbicort pMDI with space device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the λz after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered with spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Percentage of subjects who experienced treatment-related adverse events (AEs) after administration of single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device | From signing the informed consent form until 5-7 days post final dose (approximately 7 weeks)
  To assess the safety in terms of percentage of subjects who experienced treatment-related AEs after administration of single doses of budesonide and formoterol delivered via Symbicort pMDI with spacer device and with and without charcoal to healthy subjects.
  The analysis was done on the safety analysis set population which included all subjects who received at least 1 dose of Symbicort pMDI and for whom any safety post-dose data were available.
AUC after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the AUC after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
tmax after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the tmax after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
t½,λz after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the t½,λz after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Vz/F after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the Vz/F after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
CL/F after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the CL/F after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
tlast after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the tlast after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
λz after single doses of budesonide and formoterol delivered via Symbicort pMDI without spacer device | Pre-dose and at 5, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, 18 and 24 hours after Symbicort dosing
  To characterise the λz after single doses of budesonide and formoterol delivered via Symbicort pMDI when administered without spacer device and with and without charcoal under fasted condition to healthy subjects.
  The analysis was done on pharmacokinetic analysis set population.
Percentage of subjects who experienced treatment-related AEs after administration of single dose of budesonide and formoterol delivered via Symbicort pMDI without a spacer device | From signing the informed consent form until 5-7 days post final dose (approximately 7 weeks)
  To assess the safety in terms of percentage of subjects who experienced treatment-related AEs after administration of single doses of budesonide and formoterol delivered via Symbicort pMDI without the spacer device and with and without charcoal to healthy subjects. The analysis was done on the safety analysis set population which included all subjects who received at least 1 dose of Symbicort pMDI and for whom any safety post-dose data were available.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rainard Fuhr, Dr. med, Principal Investigator — PAREXEL Early Phase Clinical Unit London, United Kingdom
Locations (1):
- Research Site, Harrow, United Kingdom

REFERENCES:
- [Background] Gillen M, Forte P, Svensson JO, Lamarca R, Burke J, Rask K, Larsdotter Nilsson U, Eckerwall G. Effect of a spacer on total systemic and lung bioavailability in healthy volunteers and in vitro performance of the Symbicort(R) (budesonide/formoterol) pressurized metered dose inhaler. Pulm Pharmacol Ther. 2018 Oct;52:7-17. doi: 10.1016/j.pupt.2018.08.001. Epub 2018 Aug 2. PMID 30077809
- See also: Redacted protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4111&filename=D589WC00001%20(229149)-Protocol%20f2.0-06Dec2016_Redacted.pdf